CLINICAL TRIAL: NCT01023529
Title: A Prospective Multicenter Study of Symptoms and QOL in Patients With Prostate and Rectal Cancers Receiving Palliative Pelvic Radiation
Brief Title: Symptoms and Quality of Life (QoL) After Palliative Pelvic Radiation of Prostate and Rectal Cancers
Acronym: PallRad1
Status: Completed | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Oslo University Hospital (Other); Sykehuset Innlandet HF (Other); Nordlandssykehuset HF (Other); University Hospital of North Norway (Other); Helse Stavanger HF (Other Government); Alesund Hospital (Other); Trondheim University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-1684(REK)
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Prostatic Neoplasms; Rectal Neoplasms
Keywords: Prostatic Neoplasms; Rectal Neoplasms; Palliative treatment; Radiotherapy; Quality of life
MeSH Terms: conditions — Prostatic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prostate cancer: Patients with incurable prostate cancer requiring palliation of symptoms from a soft-tissue pelvic tumor.
  Interventions: Radiation: Palliative pelvic soft-tissue radiation (external beam)
- Rectal Cancer: Patients with incurable rectal cancer requiring palliation of symptoms from a soft-tissue pelvic tumor.
  Interventions: Radiation: Palliative pelvic soft-tissue radiation (external beam)

INTERVENTIONS:
Radiation: Palliative pelvic soft-tissue radiation (external beam) — 3 Gy x 10-13 (range 30 - 39 Gy total)

SUMMARY:
The purpose of this study is to assess the effect of palliative pelvic radiation on symptoms and quality of life among patients with incurable prostate and rectal cancer.

DETAILED DESCRIPTION:
With the aging population, the prevalence of cancer is on the rise, leading to an increased demand for effective palliative treatment. There is little scientific information describing the effects of palliative radiotherapy among patients treated for soft-tissue tumors of the pelvis. This is a treatment that is used relatively frequently, but delivered heterogeneously since the optimum fractionation schedule has yet to be established. This study aims to define the effects of one such fractionation schedule (3Gy x 10-13) and thus, establish a foundation for future fractionation studies.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Histologically or cytologically proven adenocarcinoma of the prostate or rectosigmoid colon.
* Incurable disease (hormone-resistant in cases of prostate cancer)
* Life expectancy > 3 months
* Symptomatic soft-tissue pelvic tumor mass (primary, recurrence or metastases)
* Planned fractionated radiotherapy (3Gy x 10-13)
* Written informed consent

Exclusion criteria:

* Unable to fill out questionnaires (due to language or cognitive barriers)
* New systemic tumor-targeted treatment (hormone manipulation, chemotherapy, monoclonal antibodies, etc.) started within four weeks of baseline or during the 6 weeks immediately following pelvic radiotherapy.
* Previous pelvic radiotherapy
* The presence of a second primary pelvic cancer or other cancer requiring treatment
* Currently receiving treatment with an investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic patients referred for palliative pelvic radiotherapy of prostate and rectosigmoid cancers.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2009-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Effect on patient's target symptom. | at end of treatment and 6 weeks and 12 weeks after treatment completion

SECONDARY OUTCOMES:
Effect on patient's QoL. | at end of treatment and 6 and 12 weeks after treatment completion.
Time to improvement in patient's symptoms and QoL. | at end of treatment and 6 and 12 weeks after treatment completion.

CONTACTS AND LOCATIONS:
Locations (8):
- Norway (8):
  - Stavanger University Hospital, Stavanger, Rogaland
  - Ålesund Hospital, Ålesund
  - Nordland Hospital, Bodø, Bodø
  - Innlandet Hospital Trust, Gjøvik, Gjøvik
  - Center for Cancer Treatment, Sorlandet Hospital HF, Kristiansand
  - The Cancer Center, Ullevål University Hospital, Oslo
  - University Hospital of Northern Norway (Tromsø), Tromsø
  - St. Olav's Hospital, Trondheim